CLINICAL TRIAL: NCT05245123
Title: Psychosocial Situation of Children With Rare Solid Abdominal Tumors and Their Families
Acronym: PsyRareCare
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Boettcher, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 2021-100605-BO-ff
Record Dates: First submitted 2022-01-28; First posted 2022-02-17 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Neuroblastoma; Nephroblastoma; Hepatoblastoma
Keywords: rare diseases
MeSH Terms: conditions — Neuroblastoma; Wilms Tumor; Hepatoblastoma; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Families of rare diseased children: Clinical study participants are patients who have sought treatment at the University Medical Center Hamburg-Eppendorf and University Medical Centre Mannheim due to the rare disease. Every family receives a comprehensive psychosocial diagnostic in the form of standardized instruments.
- Families in the comparative control group: Participants in the healthy control sample are matched to the clinical sample in terms of age and gender. Included are families of children aged 0-17 years, who have undergone a surgical procedure in the first 3 years of life that does not cause chronic complaints; such as hernia surgery or testicular relocation.

SUMMARY:
Families of children with rare diseases (i.e., not more than 5 out of 10.000 people are affected) are often highly burdened with fears, insecurities and concerns regarding the affected child and his/her siblings. The aim of the present research project is to examine the psychosocial burden of the children with rare solid abdominal tumors and their family in order to draw attention to a possible psychosocial care gap in this population.

DETAILED DESCRIPTION:
The central objective of the cross-sectional study is to show the psychosocial supply gap for families with children and adolescents affected by rare diseases in the field of oncology pediatric surgery. Among the rare diseases that are included are rare solid abdominal tumors. In order to have a comparative sample, additional data of a matched control group are collected. Central standardized psychosocial outcomes will be assessed from the perspectives of the parents and the affected child.

ELIGIBILITY:
Inclusion Criteria (families of rare disease):

* Family with at least one child between 0 and 17 years with rare solid abdominal tumors.
* Consent to participate in the study.
* Sufficient knowledge of the German language of parents and children.

Exclusion Criteria (families of rare disease):

- Severe acute physical, mental and/or cognitive impairment of the child, so that the questionnaire survey does not appear possible and/or unreasonable at this stage.

Inclusion Criteria (control group):

* Family with at least one child between 0 and 17 years who have undergone a surgical procedure in the first 3 years of life that does not cause chronic complaints
* Consent to participate in the study.
* Sufficient knowledge of the German language of parents and children.

Exclusion Criteria (control group):

- Families of children with a congenital or chronic disease.

Ages: 1 Month to 17 Years | Sex: All
Age Groups: Child
Study Population: Clinical study participants for the diagnostic study are patients who have sought treatment at the University Medical Center Hamburg-Eppendorf and University Medical Center Mannheim due to a rare pediatric disease. Participants in the healthy control sample are matched to the clinical sample in terms of age and gender. Included are families of children aged 0-17 years, who have undergone a surgical procedure at the University Medical Center Hamburg-Eppendorfin and University Medical Center Mannheim the first 3 years of life that does not cause chronic complaints; such as hernia surgery or testicular relocation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life of the parents (EQ-5D) | 1 minutes
  Quality of Life (QoL) of the parents, assessed from the perspective of the parents by the instrument "European Quality of Life Five Dimension" (EQ-5D; Hinz et al., 2006). The instrument consists of 5 dimensions, which are answered on a three-point scale. Higher scores indicate greater QoL.
Health-related Quality of Life of the parents (SF-12) | 4 minutes
  Health-related Quality of Life (HRQoL) of the parents, assessed from the perspective of the parents by the "Short-Form-12" (SF-12; Morfeld, Kirchberger & Bullinger, 2011). The instrument consists of 12 items. Higher scores indicate greater HRQoL.
Severity of depression (PHQ-9) | 2 minutes
  Severity of depression, will be assessed with the 9-question Patient Health Questionnaire (PHQ-9; Löwe et al., 2015). The instrument consists of 9 items. Higher scores indicate greater depression levels.
Severity of generalized anxiety disorder | 1 minutes
  Generalizied Anxiety Disorder Scale-7 (GAD-7; Spitzer, Kroenke & Löwe, 2006). The instrument consists of 7 items. Higher score indicate greater anxiety levels.
Mental health of the parents (BSI-18) | 4 minutes
  Mental health of the parents, assessed from the perspective of the parents by the "Brief Symptom Inventory-18" (BSI-18; Spitzer et al., 2011). The instrument consists of 18 items, which are answered on a five-point Likert scale (0 to 4). Higher BSI scores indicate greater psychological distress.
Health-related quality of life of the chronically-ill children/adolescents (Peds-QL 4.0) | 4 minutes
  Health-related quality of life of the chronically-ill children/adolescents, assessed from the perspective of the child/adolescent (from 10 years of age) and from the perspective of the parents by the "Pediatric Quality of Life Inventory 4.0" (Peds-QL 4.0; (Varni, Seid, & Kurtin, 2001). Items will be linearly transformed to a scale of 0 to 100, with higher scores indicating better HRQoL.
Psychiatric disorders of the chronically-ill children/adolescents (SDQ) | 4 minutes
  Psychiatric disorders of the chronically-ill children/adolescents assessed perspective of the child/adolescent and from the perspective of the parents by the "Strengths and Difficulties Questionnaire" (SDQ; Klasen, Woerner, Rothenberger, & Goodman, 2003). Items are rated on a three-point Likert scale (0 to 2). Higher scores represent greater psychopathology or greater prosocial behavior.

SECONDARY OUTCOMES:
Social support of the parents, of the chronically-ill children/adolescents (OSSS) | 3 minutes
  Social support of the parents, of the chronically-ill children/adolescents and of the siblings, assessed from the perspective of the parents, of the chronically-ill children/adolescents and from the sibling, respectively, by the "Oslo Social Support Scale" (OSSS; Dalgard, 2006). The sum score ranges from 3 to 14. The higher the sum score, the stronger the social support
Coping of the parents (CHIP-D) | 3 minutes
  Coping of the parents, assessed from the perspective of the parents by the German version of the "Coping Health Inventory for Parents" (CHIP-D; McCubbin, McCubbin, Cauble & Goldbeck, 2001). Items are rated on a four-point Likert scale (0 to 3). Higher scores represent greater use of the respective coping pattern.
Family relationships, family dynamics and functionality (FB-A) | 3 minutes
  Family relationships, family dynamics and functionality, assessed from the perspective of the parents, of the chronically-ill children/adolescents and from the sibling, respectively by "Familienbögen" (FB-A; Cierpka & Frevert, 1994). Items are rated on a four-point Likert scale (0 to 3)
Familial predispositions (FaBel) | 3 minutes
  familial predispositions assessed from the perspective of the parents by the "Familien-Belastungs-Fragebogen" (FaBel; Ravens-Sieberer, 2001). Items are rated on a four-point Likert scale ranging from 1 (is not right at all) to 4 (is completely right).
Satisfaction with the relationship and parenting relationship of the parents (PFB) | 4 minutes
  Satisfaction with the relationship and parenting relationship of the parents, assessed from the perspective of the parents by the "Partnerschaftsfragebogen" (PFB; Hahlweg, 2016).
Parent-child communication (PACS) | 4 minutes
  Parent-child communication was assessed from the perspective of the child/adolescent and from the perspective of the parents by the "Parent-Adolescent Communication Scale" (PACS; Barnes & Olsen, 1982). Items are rated on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Center Mannheim, Mannheim, Baden-Wurttemberg
  - University Medical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided